CLINICAL TRIAL: NCT05652218
Title: REsynchronization Comparison In LBBB and Normal or Mildly Reduced VENTricular Function With CRT (REINVENT-CRT), a Phase I Prospective Randomized Controlled Trial
Brief Title: REsynchronization Comparison In LBBB and Normal or Mildly Reduced VENTricular Function With CRT (REINVENT-CRT)
Acronym: REINVENT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: U22-04-4739
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-06

CONDITIONS: Left Ventricular Ejection Fraction; Heart Failure (HF); Left Bundle-Branch Block
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Intervention Model Description: single arm crossover study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Sequence 1 (Experimental): LB-CRT - Left Bundle Cardiac Resynchronization Therapy, Participants will spend 3 months in this group
  Interventions: Device: LB-CRT; Device: BIV-CRT
- Sequence 2 (Experimental): BiV-CRT - Biventricular Pacing Cardiac Resynchronization Therapy. Participants will spend 3 months in this group
  Interventions: Device: LB-CRT; Device: BIV-CRT

INTERVENTIONS:
Device: LB-CRT — LB-CRT (DDD 60-130, LV lead turned off) (active intervention #1)
Device: BIV-CRT — BIV-CRT (DDD 60- 130, LV lead turned on) (active intervention #2).

SUMMARY:
Primary Objective - To determine if implantation of a permanent CRT pacing device (with LB-CRT, or conventional BiV-CRT with a coronary sinus LV lead) can improve electromechanical function, HF symptoms, and natriuretic peptide levels among patients with symptomatic HF, LVEF > 35%, and LBBB.

DETAILED DESCRIPTION:
This pilot study will be a multicenter randomized controlled trial involving 20 medically stable outpatients with heart failure (HF), preserved or mildly reduced LVEF (>35%), and LBBB. Patients will undergo implantation of a Medtronic Percepta CRT-P with an atrial lead, left bundle branch area pacing (LBBap) lead, and a LV lead. They will then be randomly allocated in a 1:1 fashion to usual care plus LB-CRT (DDD 60-130, LV lead turned off) (active intervention #1) or usual care plus BIV-CRT (DDD 60- 130, LV lead turned on) (active intervention #2).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent form and HIPAA Authorization.
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female aged ≥18 years
* Strict LBBB defined as QRS duration ≥130ms in women and ≥140ms in men, a QS or rS complex in V1 and V2, as well as notching or QRS slurring in mid-QRS in ≥2 contiguous leads.
* NYHA II/III, ambulatory NYHA IV, or NYHA I HF with any prior history of HF symptom decompensation requiring hospitalization, ED visit, or outpatient visit for care with IV diuretic
* LVEF >35% by clinically obtained echocardiogram overread by the study core-lab
* Demonstration of adequate echocardiographic images to allow for assessment of endpoints
* On a stable guideline directed HF medical regimen
* For females of reproductive potential: use of a highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation
* Ability to understand and the willingness to sign a written informed consent form and HIPAA Authorization.

Exclusion Criteria:

* Patients with anticipated addition or titration of HF medical therapies (ACE/ARB/ARNI, beta blocker, MRA, SGLT2 inhibitor) during the duration of the study
* Treatment with another investigational drug or other intervention within 3 months
* Current unrevascularized coronary artery disease, unstable angina, acute MI, CABG, or PCI within the past 3 months
* Significant non-functional mitral or aortic valvular disease (severe stenosis or regurgitation)
* Significant structural heart [including hypertrophic cardiomyopathy (septal thickness ≥15 mm) or infiltrative cardiomyopathy (eg. amyloid)]
* Current moderate to severe pulmonary hypertension (right ventricular systolic pressure of ≥40 mmHg)
* Oxygen dependent chronic lung disease
* Prolonged episodes of AF (>3 days or an AF burden >10%) within the preceding 3 months
* Presence of cardiac pacemaker or implantable cardioverter defibrillator
* Prior mechanical tricuspid valve replacement
* Pregnancy or lactation due to concerns about the effect of radiation from the pacemaker implantation procedure on the fetus
* Known allergic reactions to components of the pacemaker or leads
* Febrile illness within 3 days of trial enrollment
* Parents/guardians or participants who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
* Control Participant Exclusion Criteria: same

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-02-26 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial performance index (MPI) as compared to Baseline | Baseline and 3 month treatment period after each pacing mode
  Myocardial performance index (MPI), a global measure of cardiac performance is defined using tissue Doppler imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Atwater, MD, Principal Investigator — Inova Health Care Services
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Inova Health System, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No